CLINICAL TRIAL: NCT04218656
Title: DUAL Pathway Inhibition (Low-dose Rivaroxaban and Aspirin) as Compared to Aspirin Only to Improve Endothelial Function in Peripheral Artery Disease.
Brief Title: DUAL Pathway Inhibition to Improve Endothelial Function in Peripheral Artery Disease
Acronym: DUAL-PAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL2019-6036
Record Dates: First submitted 2019-12-23; First posted 2020-01-06 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-02

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Two single clinical cohorts will be studied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): 111 patients with intermittent claudication
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet
- Group B (Experimental): 48 patients with critical limb ischemia with pain at rest and/or foot ulcers
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet

INTERVENTIONS:
Drug: Rivaroxaban 2.5 Mg Oral Tablet — 2.5 mg rivaroxaban twice a day in addition to Aspirin 100mg once a day (standard care).
  Other Names: Xarelto

SUMMARY:
Peripheral artery disease (PAD) is a manifestation of systemic atherosclerosis, causing patients to be at high risk of major adverse cardiovascular and limb events. Therefore, single antiplatelet therapy is recommended when patients are symptomatic or have undergone revascularization. Rivaroxaban (2.5 mg twice a day) in addition to Aspirin (100 mg once a day) has shown to be effective in reducing morbidity and mortality from major cardiovascular and limb events in patients with stable peripheral or carotid artery disease compared to Aspirin alone. Although a higher rate of major bleeding was detected, the incidence of fatal or critical organ bleedings was not increased.

Endothelial dysfunction is one of the first signs of atherosclerosis and is related to major cardiovascular events. The level of vascular endothelial dysfunction can be measured using the carotid artery reactivity (CAR) test. The investigators hypothesized that a combination of low-dose rivaroxaban and antiplatelet therapy would improve endothelial function in PAD patients.

The investigators aim to study the effectiveness of this combination therapy in improving vascular endothelial function in patients with stable or symptomatic PAD.

Therefore the investigators will study two clinical cohorts of lower extremity PAD patients (n=159) with intermittent claudication (group A: Fontaine stages 1-2) or critical limb ischemia with pain at rest and/or foot ulcers (group B: Fontaine stages 3-4) who have an indication for single antiplatelet therapy.

Aspirin 100mg once a day + 2.5 mg rivaroxaban twice a day will be given during 3 months, preceded by a run-in period of Aspirin alone (100 mg once a day) as reference.

The change in proportion of patients with CAR-constriction from baseline (Aspirin alone) to 3 months after adding low dose rivaroxaban will be compared for both study groups (A and B).

DETAILED DESCRIPTION:
Rationale: Peripheral artery disease (PAD) is a manifestation of systemic atherosclerosis, causing patients to be at high risk of major adverse cardiovascular events and major adverse limb events, including amputation. Therefore, clopidogrel or Aspirin depending on national guidelines, is recommended as single antiplatelet therapy when patients are symptomatic or have undergone revascularization. Anticoagulant therapies have not shown to be superior in PAD patients and have high rates of major bleedings. However, rivaroxaban (2.5 mg twice a day), an oral factor Xa inhibitor, in addition to Aspirin (100 mg once a day) has shown to be effective in reducing morbidity and mortality from coronary artery disease and major cardiovascular and limb events in patients with stable peripheral or carotid artery disease compared to Aspirin alone. Although a higher rate of major bleeding was detected, the incidence of fatal or critical organ bleedings was not increased.

Endothelial dysfunction is one of the first signs of atherosclerosis and is present before clinical symptoms appear. Endothelial dysfunction contributes to the progression of atherosclerosis and is related to major cardiovascular events. The level of vascular endothelial dysfunction can be measured using the carotid artery reactivity (CAR) test. This test measures the CAR in response to sympathic stimulation and can also be used to measure endothelial dysfunction in PAD patients and how a combination of rivaroxaban and Aspirin affects it. The investigators hypothesized that a combination of low-dose rivaroxaban and antiplatelet therapy would improve endothelial function in PAD patients.

Objective: To study the effectiveness of low-dose rivaroxaban with Aspirin in improving endothelial function in patients with stable or symptomatic PAD.

Study design: Two clinical cohort studies will be performed. Study population: Lower extremity PAD patients (n=159) with intermittent claudication (group A: Fontaine stages 1-2) or critical limb ischemia with pain at rest and/or foot ulcers (group B: Fontaine stages 3-4) who have an indication for single antiplatelet therapy are eligible for this study.

Intervention (if applicable): Aspirin 100mg once a day + 2.5 mg rivaroxaban twice a day (combination therapy). The use of Aspirin alone (100 mg once a day) during the run-in period is used as reference.

Main study parameters/endpoints: The primary outcome measure is the CAR after 3 months combination treatment. The change in proportion of patients with CAR-constriction from baseline (Aspirin alone) to 3 months after adding low dose rivaroxaban will be compared for both study groups (A and B). Serum endothelin-1 levels will be quantified as a marker for cardiovascular disease at baseline and 3 months after adding low dose rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic or stable lower extremity PAD patients (Fontaine stages 2-4) with an indication for single antiplatelet therapy according to international (ESC) guidelines
* >16 years old
* Written informed consent

Exclusion Criteria:

* Patients having or at risk of major bleeding:

  * Gastrointestinal ulceration
  * Current malignant neoplasms
  * Brain or spinal injury
  * Brain, spinal or ophthalmic surgery
  * Intracranial hemorrhage
  * Known or suspected esophageal varices
  * Arteriovenous malformations
  * Major intraspinal or intracerebral vascular abnormalities
  * Hepatic disease associated with coagulopathy and clinically relevant bleeding risk, including cirrhotic patients with Child Pugh B and C
  * Use of selective serotonin reuptake inhibitors or serotonin-norepinephrine reuptake inhibitors
* Patients with prosthetic valves
* Patients with a history of asthma attacks caused by salicylates
* Severe renal impairment (creatinine clearance <30 ml/min)
* Systemic treatment with strong CYP3A4 and/or P-glycoprotein inhibitors (i.e. azole-antimyotics, HIV protease inhibitors)
* Concomitant treatment with other anticoagulants
* Concomitant treatment with methotrexate at a weekly dosage of >15 mg
* Pregnant or lactating
* Known hypersensitivity to Aspirin or rivaroxaban

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Carotid artery reactivity | 3 months
  The change in proportion of patients with carotid artery reactivity constriction from baseline (Aspirin alone) to 3 months after adding low dose rivaroxaban

SECONDARY OUTCOMES:
Plasma endothelin-1 levels | 3 months
  The change in plasma endothelin-1 level as quantified by Enzyme-Linked Immuno Sorbent Assay from baseline (Aspirin alone) to 3 months after adding low-dose rivaroxaban

CONTACTS AND LOCATIONS:
Overall Officials: Michiel C Warlé, PhD, Principal Investigator — Radboud University Medical Center; Michel MPJ Reijnen, Professor, Principal Investigator — Rijnstate
Locations (2):
- Netherlands (2):
  - Rijnstate hospital, Arnhem
  - Radboudumc, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steg PG, Bhatt DL, Wilson PW, D'Agostino R Sr, Ohman EM, Rother J, Liau CS, Hirsch AT, Mas JL, Ikeda Y, Pencina MJ, Goto S; REACH Registry Investigators. One-year cardiovascular event rates in outpatients with atherothrombosis. JAMA. 2007 Mar 21;297(11):1197-206. doi: 10.1001/jama.297.11.1197. PMID 17374814
- [Background] Bhatt DL, Eagle KA, Ohman EM, Hirsch AT, Goto S, Mahoney EM, Wilson PW, Alberts MJ, D'Agostino R, Liau CS, Mas JL, Rother J, Smith SC Jr, Salette G, Contant CF, Massaro JM, Steg PG; REACH Registry Investigators. Comparative determinants of 4-year cardiovascular event rates in stable outpatients at risk of or with atherothrombosis. JAMA. 2010 Sep 22;304(12):1350-7. doi: 10.1001/jama.2010.1322. Epub 2010 Aug 30. PMID 20805624
- [Background] Brott TG, Halperin JL, Abbara S, Bacharach JM, Barr JD, Bush RL, Cates CU, Creager MA, Fowler SB, Friday G, Hertzberg VS, McIff EB, Moore WS, Panagos PD, Riles TS, Rosenwasser RH, Taylor AJ, Jacobs AK, Smith SC Jr, Anderson JL, Adams CD, Albert N, Buller CE, Creager MA, Ettinger SM, Guyton RA, Halperin JL, Hochman JS, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura RA, Ohman EM, Page RL, Riegel B, Stevenson WG, Tarkington LG, Yancy CW. 2011 ASA/ACCF/AHA/AANN/AANS/ACR/ASNR/CNS/SAIP/SCAI/SIR/SNIS/SVM/SVS guideline on the management of patients with extracranial carotid and vertebral artery disease: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines, and the American Stroke Association, American Association of Neuroscience Nurses, American Association of Neurological Surgeons, American College of Radiology, American Society of Neuroradiology, Congress of Neurological Surgeons, Society of Atherosclerosis Imaging and Prevention, Society for Cardiovascular Angiography and Interventions, Society of Interventional Radiology, Society of NeuroInterventional Surgery, Society for Vascular Medicine, and Society for Vascular Surgery. Developed in collaboration with the American Academy of Neurology and Society of Cardiovascular Computed Tomography. Catheter Cardiovasc Interv. 2013 Jan 1;81(1):E76-123. doi: 10.1002/ccd.22983. Epub 2011 Feb 3. No abstract available. PMID 23281092
- [Background] Writing Committee Members; Gerhard-Herman MD, Gornik HL, Barrett C, Barshes NR, Corriere MA, Drachman DE, Fleisher LA, Fowkes FGR, Hamburg NM, Kinlay S, Lookstein R, Misra S, Mureebe L, Olin JW, Patel RAG, Regensteiner JG, Schanzer A, Shishehbor MH, Stewart KJ, Treat-Jacobson D, Walsh ME; ACC/AHA Task Force Members; Halperin JL, Levine GN, Al-Khatib SM, Birtcher KK, Bozkurt B, Brindis RG, Cigarroa JE, Curtis LH, Fleisher LA, Gentile F, Gidding S, Hlatky MA, Ikonomidis J, Joglar J, Pressler SJ, Wijeysundera DN. 2016 AHA/ACC Guideline on the Management of Patients with Lower Extremity Peripheral Artery Disease: Executive Summary. Vasc Med. 2017 Jun;22(3):NP1-NP43. doi: 10.1177/1358863X17701592. No abstract available. PMID 28494710
- [Background] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debus S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylor AR, Roffi M, Rother J, Sprynger M, Tendera M, Tepe G, Venermo M, Vlachopoulos C, Desormais I; ESC Scientific Document Group. 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS): Document covering atherosclerotic disease of extracranial carotid and vertebral, mesenteric, renal, upper and lower extremity arteriesEndorsed by: the European Stroke Organization (ESO)The Task Force for the Diagnosis and Treatment of Peripheral Arterial Diseases of the European Society of Cardiology (ESC) and of the European Society for Vascular Surgery (ESVS). Eur Heart J. 2018 Mar 1;39(9):763-816. doi: 10.1093/eurheartj/ehx095. No abstract available. PMID 28886620
- [Background] Warfarin Antiplatelet Vascular Evaluation Trial Investigators; Anand S, Yusuf S, Xie C, Pogue J, Eikelboom J, Budaj A, Sussex B, Liu L, Guzman R, Cina C, Crowell R, Keltai M, Gosselin G. Oral anticoagulant and antiplatelet therapy and peripheral arterial disease. N Engl J Med. 2007 Jul 19;357(3):217-27. doi: 10.1056/NEJMoa065959. PMID 17634457
- [Background] Prins MH, Lensing AW, Brighton TA, Lyons RM, Rehm J, Trajanovic M, Davidson BL, Beyer-Westendorf J, Pap AF, Berkowitz SD, Cohen AT, Kovacs MJ, Wells PS, Prandoni P. Oral rivaroxaban versus enoxaparin with vitamin K antagonist for the treatment of symptomatic venous thromboembolism in patients with cancer (EINSTEIN-DVT and EINSTEIN-PE): a pooled subgroup analysis of two randomised controlled trials. Lancet Haematol. 2014 Oct;1(1):e37-46. doi: 10.1016/S2352-3026(14)70018-3. Epub 2014 Sep 28. PMID 27030066
- [Background] Mega JL, Braunwald E, Wiviott SD, Bassand JP, Bhatt DL, Bode C, Burton P, Cohen M, Cook-Bruns N, Fox KA, Goto S, Murphy SA, Plotnikov AN, Schneider D, Sun X, Verheugt FW, Gibson CM; ATLAS ACS 2-TIMI 51 Investigators. Rivaroxaban in patients with a recent acute coronary syndrome. N Engl J Med. 2012 Jan 5;366(1):9-19. doi: 10.1056/NEJMoa1112277. Epub 2011 Nov 13. PMID 22077192
- [Background] Eikelboom JW, Connolly SJ, Bosch J, Dagenais GR, Hart RG, Shestakovska O, Diaz R, Alings M, Lonn EM, Anand SS, Widimsky P, Hori M, Avezum A, Piegas LS, Branch KRH, Probstfield J, Bhatt DL, Zhu J, Liang Y, Maggioni AP, Lopez-Jaramillo P, O'Donnell M, Kakkar AK, Fox KAA, Parkhomenko AN, Ertl G, Stork S, Keltai M, Ryden L, Pogosova N, Dans AL, Lanas F, Commerford PJ, Torp-Pedersen C, Guzik TJ, Verhamme PB, Vinereanu D, Kim JH, Tonkin AM, Lewis BS, Felix C, Yusoff K, Steg PG, Metsarinne KP, Cook Bruns N, Misselwitz F, Chen E, Leong D, Yusuf S; COMPASS Investigators. Rivaroxaban with or without Aspirin in Stable Cardiovascular Disease. N Engl J Med. 2017 Oct 5;377(14):1319-1330. doi: 10.1056/NEJMoa1709118. Epub 2017 Aug 27. PMID 28844192
- [Background] Anand SS, Bosch J, Eikelboom JW, Connolly SJ, Diaz R, Widimsky P, Aboyans V, Alings M, Kakkar AK, Keltai K, Maggioni AP, Lewis BS, Stork S, Zhu J, Lopez-Jaramillo P, O'Donnell M, Commerford PJ, Vinereanu D, Pogosova N, Ryden L, Fox KAA, Bhatt DL, Misselwitz F, Varigos JD, Vanassche T, Avezum AA, Chen E, Branch K, Leong DP, Bangdiwala SI, Hart RG, Yusuf S; COMPASS Investigators. Rivaroxaban with or without aspirin in patients with stable peripheral or carotid artery disease: an international, randomised, double-blind, placebo-controlled trial. Lancet. 2018 Jan 20;391(10117):219-229. doi: 10.1016/S0140-6736(17)32409-1. Epub 2017 Nov 10. PMID 29132880
- [Background] Borissoff JI, Spronk HM, ten Cate H. The hemostatic system as a modulator of atherosclerosis. N Engl J Med. 2011 May 5;364(18):1746-60. doi: 10.1056/NEJMra1011670. No abstract available. PMID 21542745
- [Background] Spronk HM, de Jong AM, Crijns HJ, Schotten U, Van Gelder IC, Ten Cate H. Pleiotropic effects of factor Xa and thrombin: what to expect from novel anticoagulants. Cardiovasc Res. 2014 Mar 1;101(3):344-51. doi: 10.1093/cvr/cvt343. Epub 2014 Jan 2. PMID 24385341
- [Background] Esmon CT. Targeting factor Xa and thrombin: impact on coagulation and beyond. Thromb Haemost. 2014 Apr 1;111(4):625-33. doi: 10.1160/TH13-09-0730. Epub 2013 Dec 12. PMID 24336942
- [Background] Panza JA, Quyyumi AA, Brush JE Jr, Epstein SE. Abnormal endothelium-dependent vascular relaxation in patients with essential hypertension. N Engl J Med. 1990 Jul 5;323(1):22-7. doi: 10.1056/NEJM199007053230105. PMID 2355955
- [Background] Makimattila S, Virkamaki A, Groop PH, Cockcroft J, Utriainen T, Fagerudd J, Yki-Jarvinen H. Chronic hyperglycemia impairs endothelial function and insulin sensitivity via different mechanisms in insulin-dependent diabetes mellitus. Circulation. 1996 Sep 15;94(6):1276-82. doi: 10.1161/01.cir.94.6.1276. PMID 8822980
- [Background] Casino PR, Kilcoyne CM, Quyyumi AA, Hoeg JM, Panza JA. The role of nitric oxide in endothelium-dependent vasodilation of hypercholesterolemic patients. Circulation. 1993 Dec;88(6):2541-7. doi: 10.1161/01.cir.88.6.2541. PMID 8252665
- [Background] Celermajer DS, Sorensen KE, Spiegelhalter DJ, Georgakopoulos D, Robinson J, Deanfield JE. Aging is associated with endothelial dysfunction in healthy men years before the age-related decline in women. J Am Coll Cardiol. 1994 Aug;24(2):471-6. doi: 10.1016/0735-1097(94)90305-0. PMID 8034885
- [Background] Lerman A, Zeiher AM. Endothelial function: cardiac events. Circulation. 2005 Jan 25;111(3):363-8. doi: 10.1161/01.CIR.0000153339.27064.14. No abstract available. PMID 15668353
- [Background] Rubinshtein R, Kuvin JT, Soffler M, Lennon RJ, Lavi S, Nelson RE, Pumper GM, Lerman LO, Lerman A. Assessment of endothelial function by non-invasive peripheral arterial tonometry predicts late cardiovascular adverse events. Eur Heart J. 2010 May;31(9):1142-8. doi: 10.1093/eurheartj/ehq010. Epub 2010 Feb 24. PMID 20181680
- [Background] van Mil ACCM, Pouwels S, Wilbrink J, Warle MC, Thijssen DHJ. Carotid Artery Reactivity Predicts Events in Peripheral Arterial Disease Patients. Ann Surg. 2019 Apr;269(4):767-773. doi: 10.1097/SLA.0000000000002558. PMID 29064890
- [Background] Leentjens J, Bekkering S, Joosten LAB, Netea MG, Burgner DP, Riksen NP. Trained Innate Immunity as a Novel Mechanism Linking Infection and the Development of Atherosclerosis. Circ Res. 2018 Mar 2;122(5):664-669. doi: 10.1161/CIRCRESAHA.117.312465. Epub 2018 Jan 24. PMID 29367213
- [Derived] Willems LH, Thijssen DHJ, Groh LA, Kooijman NI, Ten Cate H, Spronk HMH, Donders ART, van der Vijver-Coppen RJ, van Hoek F, Nagy M, Reijnen MMPJ, Warle MC. Dual pathway inhibition as compared to acetylsalicylic acid monotherapy in relation to endothelial function in peripheral artery disease, a phase IV clinical trial. Front Cardiovasc Med. 2022 Oct 6;9:979819. doi: 10.3389/fcvm.2022.979819. eCollection 2022. PMID 36277757